CLINICAL TRIAL: NCT05305716
Title: Effects of Online Pilates Training on Pregnant Women During the COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: Online Pilates Training on Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Bulguroglu, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy; COVID-19; Pilates
Keywords: Pilates exercises; Pregnant; Depression; Anxiety
MeSH Terms: conditions — COVID-19; Depression; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online pilates group (Experimental): Online pilates training was done for a total of 8 weeks, 2 days a week for 1 hour. Microsoft Teams program was used to perform the exercises online. The investigators divided the individuals in the online pilates exercise group into seven smaller groups of 3 or 4 to verify whether they correctly did the exercises. A program including 15 minutes of warm-up, 30 minutes of Pilates exercises and 15 minutes of cooling and stretching exercises was arranged for the online pilates group and the exercises were performed as 10 repetitions. The exercise program recommended by the Australian Pilates and Physiotherapy Institute during pregnancy was used in the online training.
  Interventions: Other: Online Pilates Training
- control group (Active Comparator): The control group was given breathing and relaxation exercises, which they would do two days a week for eight weeks, in the form of a home program. Diaphragmatic breathing and respiratory control were given as breathing exercises.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Online Pilates Training — The group that received telerehabilitation and telerehabilitation-based pilates training.
  Arms: online pilates group
Other: Control group — The group who received breathing and relaxation exercises with a home program.
  Arms: control group

SUMMARY:
Studies show that pregnant women reduce their physical activity levels during pregnancy. The pandemic process causes the physical activities of pregnant women to decrease even more and causes a number of problems. This study aims to reveal effect of online Pilates exercises with a physiotherapist during the pandemic conducted on depression, anxiety and fear of childbirth levels of pregnant women. A total of 50 volunteer pregnant women, 26 online pilates group (OPG) and 24 control group (CG), who met the inclusion criteria of the study, were included in our study randomly. The OPG was given online Pilates exercises by the physiotherapist in groups 2 days a week for 8 weeks, 1 h a day. The CG was given a home program consisting of relaxation and breathing exercises. Depression levels; with the Edinburgh Postpartum Depression Scale, anxiety; with the State-Trait Anxiety Inventory, fear of childbirth; with the Wijma Birth Expectation/Experience Scale version B were evaluated before and after the study by using the online questionnaire form filling method. As a result of the online pilates training, there was an improvement in the all test scores (p<0.05), while no change was observed in the control group (p>0.05). In the light of these results, 8-week online pilates training applied to gain a healthy habit during the pandemic process and increase physical activity levels of the pregnant women has been concluded to be effective in reducing the levels of depression, anxiety and fear of childbirth.

DETAILED DESCRIPTION:
Although there are studies investigating the effectiveness of telerehabilitation in the literature, no online study has been found on pregnancy. The pandemic process reduces the rate of participation of pregnant women in face-to-face exercises, causing physical activity levels to decrease further. Therefore, there is a need for studies on the pregnancy process in the field of telerehabilitation. This study aims to understand how the depression, anxiety and fear of childbirth levels of pregnant women who do pilates online with a physiotherapist during the pandemic process and to bring a new approach to the field of tele-rehabilitation.

The investigators conducted the study at Ankara Medipol University, Faculty of Health Sciences, Department of Physical Therapy and Rehabilitation. This study was conducted by the principles set out in the Declaration of Helsinki. Fifty-three pregnant women aged 20-35, who completed the first trimester and had a single baby pregnancy, were included in the study, conducted under a specialist obstetrician's guidance. The exclusion criteria for this study were: multiple pregnancies; history of cardiovascular diseases, medical complications (hemorrhage, preeclampsia, placenta previa etc.) and/or cognitive disorders; contraindication for physical exercise (eg: having severe other musculoskeletal disease, high risk pregnancies, balance deficiencies); and participating in other exercises or physiotherapy programs.

* Procedures The investigators assessed the participants by an experienced physiotherapist, who was blind to the randomization, at the start of the study and after the 8-week training. The group on which they depended was not disclosed to the participants until the end of the baseline evaluation. The investigators used a computer program for randomization and randomly placed individuals who completed the initial assessment into the online pilates group (OPG) or control group (CG). The investigators performed the Pilates exercises online, under the supervision of a certified physiotherapist with 10 years of experience. The investigators asked the individuals not to inform the evaluator of their involvement in the training during the last evaluation. Before the study, the investigators explained the purpose and content of the study to the participants and obtained written informed consent from all pregnant women to participate in the study.
* Intervention Online pilates training was done by an Australian Pilates and Physiotherapy Institute certified and experienced Ph.D. Physiotherapist Halil Ibrahim Bulguroglu lasted a total of 8 weeks, 2 days a week for 1 h. Microsoft Teams program was used to perform the exercises online. The investigators divided the individuals in the Pilates exercise group into seven smaller groups of 3 or 4 to verify whether they correctly did the exercises. In this study, the investigators organized a program to include 15 min of warm-up, 30 min of Pilates exercises, and 15 min of cooling and stretching exercises, and the exercises were done in 10 repetitions. The exercise program recommended by the Australian Pilates and Physiotherapy Institute during pregnancy was used in the training. During the Pilates exercises, investigators described the exercises with different visual simulation techniques, and exercises were done together with Pilates breathing. The intensity of the exercises was increased by using different positions and elastic bands. The resistance was increased by starting with the red Therabant and switching to the blue band after two weeks. If the new resistance amount was challenging for the patient, the exercises were continued with the same color band for one more week. Stretching exercises and posture exercises were used during the cooling period. The subjects in the online pilates group were informed about side effects such as shortness of breath, dizziness, headache, muscle pain, and weakness. They were asked to stop exercising when there were any side effects.

The control group was given breathing and relaxation exercises, which they would do two days a week for eight weeks, in the form of a home program. Diaphragmatic breathing and respiratory control were given as breathing exercises.

It was stated that after the study was completed, pregnant women in the control group could also participate in the online exercise program. 6 pregnant women in the control group participated in the online pilates program after the study.

* Outcome measurements The pregnant women included in the study were evaluated with data collection forms filled with an online questionnaire twice, before and after the training programs. The investigators recorded demographic information (age, body weight, height, body mass index) of the participants.

The investigators evaluated depression with the Edinburgh Postpartum Depression Scale (EPDS). In a study conducted in 2009, it was reported that EPDS is a reliable tool in the evaluation of depressive symptoms in pregnancy. EPDS is a self-report scale consisting of 10 items, in a 4-point Likert format. The lowest score that can be obtained from the scale is 0, and the highest score is 30. The cut-off point for EPDS is 13 points. Accordingly, 13 points and above indicate the risk of depression.

The investigators assessed anxiety with the State-Trait Anxiety Inventory (STAI Form 1-2). The scale is a Likert-type scale consisting of 20 questions that measure state and trait anxiety levels separately. There are two kinds of expressions in the scales. These are called direct and reverse expressions. Direct expressions, negative emotions; reversed expressions express positive emotions. The scores obtained from both scales separately vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.

The investigators evaluated Fear of Birth with the Wijma Birth expectation/Experience Questionnaire (W-DEQ). The W-DEQ was developed to measure the nature of the fear of childbirth during and after labor by asking women questions about their expectations before birth (version A) and their experiences after birth (version B).

Data availability The data associated with the paper are not publicly available but are available from the corresponding author on reasonable request.

* Statistical analysis The investigators performed statistical analysis by using SPSS software, version 21 (SPSS Inc. Chicago, IL, USA). The normal distribution of variables was determined using histograms, probability plots, and a Shapiro-Wilk test. Because of an abnormal distribution, median and interquartile range (IQR) were used for descriptive statistics. Numerical variables showing normal distribution were shown as mean±standard deviation. The investigators used a Mann-Whitney U test to compare baseline and change values between groups. The investigators used Wilcoxon Test for comparing baseline values within the group and values after 8 weeks. The level of significance was set at p < 0.05 for all analyses. The effect sizes were evaluated according to Cohen's d standards within the pre-post differences. Effect size results were interpreted as small (≥ 0.2), medium (≥ 0.5), or large (≥ 0.8) according to guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 years of age
* Voluntarily participate in research to accept
* 12-28 weeks of pregnancy
* Singleton pregnancy

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, hearing, and perception problems that may affect the results of the research.
* Participating in other exercises or physiotherapy programs during the past 6 months.
* Multiple pregnancies

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Depression- Baseline | Assessment will be conducted before the intervention
  Edinburgh Postpartum Depression Scale (EPDS) is a self-report scale consisting of 10 items, in a 4-point Likert format. The lowest score that can be obtained from the scale is 0, and the highest score is 30. The cut-off point for EPDS is 13 points. Accordingly, 13 points and above indicate the risk of depression.
Depression-Post intervention | Assessment will be conducted immediately after the intervention
  Edinburgh Postpartum Depression Scale (EPDS) is a self-report scale consisting of 10 items, in a 4-point Likert format. The lowest score that can be obtained from the scale is 0, and the highest score is 30. The cut-off point for EPDS is 13 points. Accordingly, 13 points and above indicate the risk of depression.
Anxiety- Baseline | Assessment will be conducted before the intervention
  State-Trait Anxiety Inventory is a Likert-type scale consisting of 20 questions that measures state and trait anxiety levels separately. There are two kinds of expressions in the scales. These are called direct and reverse expressions. Direct expressions, negative emotions; reversed expressions express positive emotions. The scores obtained from both scales separately vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Anxiety-Post intervention | Assessment will be conducted immediately after the intervention
  State-Trait Anxiety Inventory is a Likert-type scale consisting of 20 questions that measures state and trait anxiety levels separately. There are two kinds of expressions in the scales. These are called direct and reverse expressions. Direct expressions, negative emotions; reversed expressions express positive emotions. The scores obtained from both scales separately vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Fear of Childbirth- Baseline | Assessment will be conducted before the intervention
  The Wijma Birth Expectation/Experience Scale version B was developed to measure the nature of the fear of childbirth during and after labor by asking women questions about their experiences after birth. The minimum score on the scale is 33, the maximum score is 198.
Fear of Childbirth-Post intervention | Assessment will be conducted immediately after the intervention
  The Wijma Birth Expectation/Experience Scale version B was developed to measure the nature of the fear of childbirth during and after labor by asking women questions about their experiences after birth. The minimum score on the scale is 33, the maximum score is 198

CONTACTS AND LOCATIONS:
Overall Officials: HALIL IB BULGUROGLU, PHD PT, Principal Investigator — Ankara Medipol University
Locations (1):
- Ankara Medipol University, Altındağ, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Arundell L, Salmon J, Timperio A, Sahlqvist S, Uddin R, Veitch J, Ridgers ND, Brown H, Parker K. Physical activity and active recreation before and during COVID-19: The Our Life at Home study. J Sci Med Sport. 2022 Mar;25(3):235-241. doi: 10.1016/j.jsams.2021.10.004. Epub 2021 Oct 14. PMID 34742627
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Bunevicius A, Kusminskas L, Pop VJ, Pedersen CA, Bunevicius R. Screening for antenatal depression with the Edinburgh Depression Scale. J Psychosom Obstet Gynaecol. 2009 Dec;30(4):238-43. doi: 10.3109/01674820903230708. PMID 19845492
- [Background] Wijma K, Wijma B, Zar M. Psychometric aspects of the W-DEQ; a new questionnaire for the measurement of fear of childbirth. J Psychosom Obstet Gynaecol. 1998 Jun;19(2):84-97. doi: 10.3109/01674829809048501. PMID 9638601
- [Result] Suner-Keklik S, Numanoglu-Akbas A, Cobanoglu G, Kafa N, Guzel NA. An online pilates exercise program is effective on proprioception and core muscle endurance in a randomized controlled trial. Ir J Med Sci. 2022 Oct;191(5):2133-2139. doi: 10.1007/s11845-021-02840-8. Epub 2021 Oct 30. PMID 34716884
- [Derived] Bulguroglu M, Bulguroglu HI. The effects of online pilates on the mood and fear of birth of pregnant women: a randomized controlled study. Sci Rep. 2024 Jul 12;14(1):16143. doi: 10.1038/s41598-024-67290-5. PMID 38997441